CLINICAL TRIAL: NCT06992141
Title: CHIVAS- M1 (Controlled Human Infection for Vaccination Against Streptococcus Pyogenes M1UK): Expanding the Scope of Experimental Human Streptococcus Pyogenes Pharyngitis
Brief Title: A Strep Throat Controlled Human Infection Trial in Healthy Adults
Acronym: CHIVAS-M1
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Auckland, New Zealand (Other); University of Melbourne (Other); University of Wollongong (Other); Université Libre de Bruxelles (Other); University of California, San Diego (Other); Leducq Foundation (Other); National Health and Medical Research Council, Australia (Other); Monash University (Other); Duke University (Other); The University of Queensland (Other); Doherty Clinical Trials Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHIVAS-M1
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-05

CONDITIONS: Streptococcus Pyogenes Pharyngitis; Streptococcus Infection
Keywords: Streptococcus pyogenes; Streptococcus pyogenes pharyngitis; Controlled Human Infection Model; S. pyogenes M1UK
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Intervention Model Description: This is an observational, sequential, dose escalation/de-escalation study with 4 predetermined doses of bacteria for human challenge. The aim is to reliably and safely cause pharyngitis in greater than or equal to 60% of participants. The starting dose is based upon the successful dose from the previous human challenge study (CHIVAS- M75) and escalation/de-escalation decisions will be based upon the number of participants diagnosed with pharyngitis in each cohort of 10-20 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human challenge participants (Experimental): Participants will be allocated a dose of M1 S. pyogenes sequentially by date of challenge based on the attack rate in the preceding participants. Up to 4 dose levels will be tested commencing at 1-5 x10^5 CFU/mL, increasing by 1 log to a maximum dose of 1-5 x 10^7 CFU/mL, or decreasing by 1 log to a minimum dose of 1-5 x 10^4 CFU/mL.
  Interventions: Biological: Streptococcus pyogenes M1UK strain MCRI0102

INTERVENTIONS:
Biological: Streptococcus pyogenes M1UK strain MCRI0102 — Human challenge with S. pyogenes M1UK strain MCRI0102

SUMMARY:
This aim of this study is to further develop a new way to study the bacteria that causes pharyngitis (strep throat). The scientific name for this bacterium is Streptococcus pyogenes and it is commonly known as Strep A. Strep A is a common type of bacteria that can cause various infections. These range from skin infections and strep throat to more serious conditions like rheumatic heart disease. In recent years there has been an increase in severe Strep A infections in most countries. Many of these cases have been reported in the news.

Human challenge models are studies which allow researchers to study organisms that cause infections in humans. In this human challenge model study, healthy participants will be carefully exposed to a specific type of Strep A under controlled conditions to cause sore throat and learn more about how Strep A causes infection. The study team has already developed a safe human challenge model using a strain of Strep A called M75. This study will use a different strain of Strep A, called M1.

The main goal of this study is to check if the procedure is safe for participants and to understand how the participant's body responds to M1 Strep A. The study will explore:

1. How much M1 Strep A is required to cause an infection.
2. How M1 Strep A grows in the body.
3. How the body reacts to M1 Strep A.

The information the investigators will get about M1 Strep A from this study will help plan future research. It may also help in designing better studies to test vaccines against Strep A.

DETAILED DESCRIPTION:
Streptococcus pyogenes infection is a major cause of death and disability globally, particularly in settings of disadvantage with a disproportionately high burden in Indigenous Australians and the Pacific region. Acute infections due to S. pyogenes range from very common superficial skin infections (>150 million prevalent cases worldwide) and pharyngitis (> 600 million incident cases) to life-threatening invasive disease (>600,000 incident cases). Post-infectious sequelae of S. pyogenes include acute rheumatic fever (ARF, ~500,000 incident cases) leading to rheumatic heart disease (RHD) (~40 million prevalent cases), and acute post-streptococcal glomerulonephritis (APSGN). The health services impact of S. pyogenes disease in all its forms is immense and strikes at every level from primary to intensive care, with associated direct and indirect costs (e.g. primary and hospital care, work and school absences, antibiotic use and misuse leading to antimicrobial resistance).

A vaccine against S. pyogenes would be a global game changer and is the only plausible way to prevent S. pyogenes infections and sequelae. Efforts to control S. pyogenes-related disease through primary prevention have proved expensive and ineffective. Animal models of S. pyogenes disease have not delivered a vaccine. S. pyogenes-related disease is an important global driver of broad-spectrum antibiotic use leading to increased antimicrobial resistance (AMR). Multiple economic analyses have shown that a vaccine against S. pyogenes would be economically viable and result in enormous healthcare savings. The World Health Organization (WHO) recognises the need for a vaccine against S. pyogenes and has prioritised vaccine development as well as adopting a resolution to end ARF and RHD at the 2018 World Health Assembly.

In the recent CHIVAS-M75 project, a diverse team of investigators developed the world's only modern S. pyogenes controlled human infection model (CHIM) using an M75 strain of S. pyogenes, following a careful and intensive approach to select and manufacture an initial challenge strain and produce a clinically relevant protocol to protect participants and maximise the model's strategic and scientific impact.

M1 strains are the leading cause of S. pyogenes infections globally and have been the principal focus of decades of 'wet' and 'dry' laboratory research that underlies current understanding of host-pathogen interactions. In 2019 a new M1 clone was described in the UK (M1UK) which has now established global dominance. M1UK is associated with outbreaks of invasive disease and scarlet fever as well as pharyngitis. Having shown the safety and reliability of human challenge using M75, an emm-type that is a relatively uncommon cause of complicated S. pyogenes disease, the M1UK strain provides a unique opportunity to study a leading emm-type associated with increasing rates of complicated S. pyogenes disease. An M1UK CHIM used in a vaccine efficacy trial could demonstrate reduced rates of pharyngitis (the most clinically relevant endpoint) that would be expected to translate to protection against invasive disease and post-streptococcal complications.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18 - 40 years (inclusive) on the day of informed consent.
2. Medically healthy, which can be determined by medical history, physical examination, BMI, transthoracic echocardiogram, non-clinically significant laboratory profiles, vital signs, and 12-lead ECG at screening, as deemed necessary by the research physician or investigator.
3. Systolic blood pressure (SBP) of 90 mmHg - 140 mmHg and diastolic blood pressure (DBP) of 60 mmHg - 90 mmHg. Vital signs can be repeated up to two times.
4. Resting heart rate (HR) of 55-100 bpm (confirmed by one repeat at screening).
5. Females must be non-pregnant, non-lactating, or postmenopausal for at least 1 year (as confirmed by follicle-stimulating hormone [FSH]), or surgically sterile for at least 6 months prior to dosing.

   Females of childbearing potential will be required to use an effective form of contraception from the time of signing informed consent until the second planned outpatient visit approximately 1 month following the inpatient challenge admission.
6. Males must not have a pregnant partner and must agree to use condoms as a method of contraception from the time of signing informed consent until the second planned outpatient visit approximately 1 month following the inpatient challenge admission.
7. Must be willing and able to read, understand, and sign the participant information and consent form. Willing to comply with all study requirements, including the inpatient period and outpatient visits for the duration of the study (approx. 3 months).
8. Willing to abstain from the use of mouthwash from the day of screening until the first outpatient visit at one week post discharge.

Exclusion Criteria:

1. History of any clinically important cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
2. Significant history of hospitalisation for illness within the six months prior to enrolment into study, or major surgery within the 12 months prior to enrolment into study, as assessed by research physician or investigator.
3. History of tonsillectomy, adenoidectomy or splenectomy.
4. Known or suspected autoimmune disease or impairment/alteration of immune function resulting from:

   1. Congenital or acquired immunodeficiency (including immunoglobulin A [IgA] deficiency)
   2. Receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
5. History of a severe drug reaction or severe allergic reaction (eg. anaphylaxis, convulsions) or clinically significant allergic disease diagnosed by a physician.
6. Personal or family history of severe S. pyogenes infection (toxic shock syndrome, necrotizing fasciitis, bloodstream infection, pleural empyema, meningitis) or post-infectious sequelae (such as acute rheumatic fever, rheumatic heart disease, post-streptococcal glomerulonephritis).
7. Clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion, e.g. gastrectomy, diarrhoea.
8. Any vaccination within the last 28 days or use of any antibiotic therapy during the 14 days before challenge.
9. Presence of an acute infectious disease or febrile illness (e.g., sub-lingual temperature ≥ 38.5°C) within the five days prior to inoculation.
10. Significant acute or chronic infection within 14 days prior to inoculation that the research physician or investigator deems may compromise participant safety.
11. Any clinically significant abnormal finding on biochemistry or haematology blood tests, urine analysis, ECG or transthoracic echocardiogram.
12. Positive serologic results for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
13. Ex-smoker with a >10 pack per year smoking history or a current smoker who is unable to stop smoking for the duration of the study.
14. History or presence of alcohol abuse (defined as regular alcohol consumption of more than 40g per day) or drug habituation, or any prior intravenous usage of an illicit substance.
15. A positive alcohol breath test at screening or admission.
16. A positive urine drug test at screening or admission (e.g., amphetamines, barbiturates, benzodiazepines, cocaine, methylenedioxymethamphetamine [MDMA], methamphetamine, methadone, opiates, phencyclidine [PCP] and tetrahydrocannabinol [THC]) unless there is an explanation acceptable to the Investigator (e.g. the participant has stated in advance that they consumed a prescription or over-the-counter product which contained the detected drug) and the participant has a negative urine drug screen on retest.
17. A positive point of care (POC) test for S. pyogenes on screening or day -1 throat swab.
18. Known hypersensitivity to more than two of the following antibiotics: penicillin, azithromycin, clindamycin, or other beta-lactam antibiotic(s).
19. Known hypersensitivity to soya protein.
20. Have participated in previous S. pyogenes challenge studies (with application of challenge agent).
21. Intolerance of throat swab procedure (exaggerated gag reflex).
22. Systemic corticosteroid in the 14 days prior to admission, or for more than seven consecutive days within the past 3 months, or anticipated use during the study period.
23. Any chronic (more than 1 month) use of inhaled high potency corticosteroids (budesonide 800 μg or fluticasone 750 μg per day).
24. Any intranasal corticosteroid use is not allowed in the 14 days prior to admission, during the inpatient period, and is discouraged prior to the first outpatient visit. Topical corticosteroid use is allowed.
25. Any use of drugs which may suppress the hypothalamic-pituitary-adrenal (HPA) axis such as adrenocorticotrophic hormone (ACTH) within the previous 3 months.
26. Any anti-inflammatory drugs (besides sporadic use of non-steroidal anti-inflammatory drugs), immunomodulators (such as monoclonal antibodies) or anticoagulants in the previous 3 months, or anticipated use of such drugs during the study period.
27. Use of prescription or non-prescription drugs and herbal supplements (such as St John´s Wort) within 14 days or 5 half-lives (whichever is the longer) prior to the inoculation administration. Use of vitamin supplements taken at standard doses is allowed.
28. Participation in a research study that involved blood sampling of more than 450 mL/1 unit of blood, received or donated blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within 3 months of informed consent.
29. History of severe infections requiring hospitalisation for intravenous antibiotics (within the last 10 years). Exceptions to this would include a short course of intravenous antibiotics for appendicitis, biliary sepsis, diverticulitis and cellulitis or a similar non-severe infection.
30. History of cancer (except adequately treated squamous cell or basal cell carcinoma of the skin and cervical intraepithelial neoplasia).
31. Presence of implants or prosthesis (e.g. artificial joints, pacemakers) deemed significant for infective complications as assessed by research physician or investigator. Participants with cosmetic implants or prosthesis may be included, as per principal investigator's discretion.
32. Participation in another research study within the 30 days prior to enrolment involving an investigational product or other intervention that might affect risk of invasive S. pyogenes infection or compromise the integrity of the study (e.g. significant volumes of blood already taken in previous study).
33. Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the results of the study, or the participant's ability to participate in the study.
34. Any employee of the sponsor or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, sibling, or child whether biological or legally adopted.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants at each dose level of M1 S. pyogenes who reach the study pharyngitis endpoint | Up to 5 days after the challenge dose of M1 S. pyogenes is administered
  The proportion of participants at each M1 S. pyogenes dose level who develop pharyngitis, using a combined clinical-microbiological definition comprising sore throat, physical examination signs of pharyngitis and tonsillitis, and microbiological confirmation of S. pyogenes by culture and nucleic acid amplification test of throat swabs

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Osowicki, FRACP PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Doherty Clinical Trials Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared by the sponsor with study collaborators upon request and as necessary to facilitate research collaborations and study publications.
  Planned sharing of de-identified IPD includes microbiological, immunologic and gene expression data gathered from study participants.
  De-identified IPD will be published in peer-reviewed journals.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified IPD will be available at the end of the clinical trial. IPD will be stored for 15 years afterwards in concordance with the International Council for Harmonisation (ICH) guidelines for clinical trial data.
Access Criteria: Only authorised study site staff will have access to source documentation. De-identified IPD will be shared with the sponsor. De-identified IPD will be shared with collaborators only in specific circumstances where sharing the data will benefit and extend research collaborations. Collaborators in this study are located in the following countries: Australian (Victoria, Queensland, Western Australia, and New South Wales), New Zealand, Belgium, Netherlands, the UK, and the US.
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre

REFERENCES:
- [Background] Osowicki J, Azzopardi KI, Fabri L, Frost HR, Rivera-Hernandez T, Neeland MR, Whitcombe AL, Grobler A, Gutman SJ, Baker C, Wong JMF, Lickliter JD, Waddington CS, Pandey M, Schuster T, Cheng AC, Pollard AJ, McCarthy JS, Good MF, Dale JB, Batzloff M, Moreland NJ, Walker MJ, Carapetis JR, Smeesters PR, Steer AC. A controlled human infection model of Streptococcus pyogenes pharyngitis (CHIVAS-M75): an observational, dose-finding study. Lancet Microbe. 2021 Jul;2(7):e291-e299. doi: 10.1016/S2666-5247(20)30240-8. Epub 2021 Apr 15. PMID 35544165